CLINICAL TRIAL: NCT05718960
Title: Randomised Trial of Traditional Dietary Advice Versus Reassurance-alone in Postprandial Functional Dyspepsia
Brief Title: Traditional Dietary Advice Versus Reassurance-alone in Postprandial Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH20655a
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dyspepsia; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reassurance-alone (Placebo Comparator)
  Interventions: Other: Reassurance-alone
- Traditional Dietary Advice (Active Comparator)
  Interventions: Behavioral: Traditional dietary advice

INTERVENTIONS:
Other: Reassurance-alone — To be informed of the absence of organic disease and provided a diagnostic explanation of functional dyspepsia
  Arms: Reassurance-alone
Behavioral: Traditional dietary advice — To receive the same information as reassurance-alone group but also recommended to eat smaller, regular meals and reduce the intake of caffeine/alcohol/fizzy drinks, fatty/processed/spicy foods, and fibre
  Arms: Traditional Dietary Advice

SUMMARY:
Functional dyspepsia is common, affecting 7.2% of the global population, and associated with substantial health impairment. Almost 80% of patients with functional dyspepsia report meal-related symptoms and are classified as having the postprandial distress syndrome (PDS) variant. However, studies evaluating dietary modifications in PDS are sparse.

The investigators will perform a single-centre randomised trial evaluating traditional dietary advice (TDA) in PDS.

50 patients with PDS will be randomly assigned to a leaflet explaining reassurance-alone +/- TDA. The reassurance-alone group will be informed of the absence of organic disease and provided a diagnostic explanation of functional dyspepsia. The TDA group will receive the same information but also be recommended to eat smaller, regular meals and reduce the intake of caffeine/alcohol/fizzy drinks, fatty/processed/spicy foods, and fibre.

Questionnaires are to be completed during the 4-week trial, including self-reported adequate relief of dyspeptic symptoms, and the validated Leuven Postprandial Distress Scale (LPDS), Gastrointestinal Symptom Rating Scale, and Napean Dyspepsia Quality of Life Index.

The primary endpoint(s) to define clinical response will be evaluated over weeks 3-4 as, i) ≥50% adequate relief of dyspeptic symptoms, and ii) >0.5-point reduction in the PDS subscale of the LPDS (calculated as the mean scores for early satiety, postprandial fullness, and upper abdominal bloating).

ELIGIBILITY:
Inclusion Criteria:

* Fulfil Rome IV symptoms criteria for functional dyspepsia
* Normal upper gastrointestinal endoscopy within last 3 years
* Online access
* English literate

Exclusion Criteria:

* Organic gastrointestinal diseases (e.g. inflammatory bowel disease, GI cancer, coeliac disease)
* Major abdominal surgery (except laparoscopy, appendectomy, cholecystectomy)
* Documented H.pylori in the last 3 months
* History of eating disorders
* Body mass index <20
* Current use of opioids or anti-inflammatory drugs
* Severe systemic disease (e.g. cardiac, renal, respiratory) necessitating frequent medical consultations
* Pregnant
* Diabetes mellitus
* Scleroderma
* Memory impairment
* Current dietary interventions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of clinical responders between traditional dietary advice vs. reassurance alone based on the leuven postprandial distress scale (LPDS) | 4 weeks
  The Leuven Postprandial Distress Scale (LPDS) assesses the severity of 8 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). A difference of 0.7 from baseline for the cardinal PDS symptoms (average of first 3 questions) will be used as a cut-off to determine clinical response by comparing averaged pre-treatment scores with the average score during the weeks 3-4.
Proportion of clinical responders between traditional dietary advice vs. reassurance alone | 4 weeks
  Self-reported adequate relief of dyspeptic symptoms as a binary answer (yes or no). A responder will be defined if ≥50% adequate relief of dyspeptic symptoms during weeks 3-4

SECONDARY OUTCOMES:
Changes in Gastrointestinal Symptom Rating Irritable Bowel syndrome Scale | 4 weeks
  The validated Gastrointestinal Symptom Rating Scale assesses the symptoms of irritable bowel syndrome, depicting problems with satiety, abdominal pain, diarrhoea, constipation and bloating. Higher scores represent greater symptom severity. Change in monthly scores will be compared within- and between-treatments for both cohorts combined.
Changes in Napean Dyspepsia-related Quality of Life Index | 4 weeks
  The Napean Dyspepsia Scale is a validated questionnaire assessing dyspepsia-related quality of life syndrome, with higher scores representing worse quality of life. Change in monthly scores will be compared within- and between-treatments for both cohorts combined.
Changes in Hospital Anxiety and Depression scale | 4 weeks
  The Hospital Anxiety and Depression Scale is a validated questionnaire assessing mood, with higher scores representing worse mood. Change in monthly scores will be compared within- and between-treatments for both cohorts combined.
Changes in Somatic Symptom reporting | 4 weeks
  The validated patient health questionnaire-12 assess extra-intestinal somatic symptoms, with higher scores representing greater somatic symptom severity. Change in monthly scores will be compared within- and between-treatments for both cohorts combined.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No